CLINICAL TRIAL: NCT00442299
Title: Phase 1 Study of Albumin Dialysis Using Prometheus in End Stage Renal Disease: Detoxification Capacity and Impact on Vascular Endothelial Function
Brief Title: Albumin Dialysis in End-Stage Renal Disease: Detoxification Capacity and Impact on Vascular Endothelial Function
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Major side-effects
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ML3041
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2007-02

CONDITIONS: Chronic Kidney Disease
Keywords: hemodialysis, urmeic retention solute, biocompatibility
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Fractionated Plasma Separation and Adsorption (FPSA)

SUMMARY:
The uremic syndrome is mainly related to the retention of a host of compounds, due to altered glomerular filtration and other factors of renal dysfunction, e.g. tubular secretion. Uremic retention solutes are arbitrarily subdivided in three different categories according to their physicochemical characteristics and their subsequent behaviour during dialysis: (i) the small, water-soluble, non-protein bound compounds, (ii) the larger middle molecules, mainly peptides and (iii) the small protein-bound compounds (1).

Although direct proof is lacking, several lines of evidence indicate that albumin is the most important carrier protein. Removal of protein bound uremic retention solutes is limited.

The Prometheus® system fractionates blood into plasma and cellular components, using an albumin-permeable polysulfon filter (AlbuFlow®) with a specially designed sieving coefficient curve (1.0 for 2-microglobulin, >0.6 for albumin, <0.3 for IgG, <0.1 for fibrinogen and <0.01 for IgM). Due to the high sieving coefficient of the filter for large molecules (i.e. cut-off at about 250 kD) molecules up to the size of albumin (69 kD) easily pass from blood into the secondary circuit which is filled with isotonic sodium chloride solution, whereas larger molecules like fibrinogen (340 kD) cannot pass through the filter. In the secondary circuit the filtered plasma with the albumin-bound toxins flows through one or two adsorbers in a row with maximized adsorption capacity for putative liver toxins that are directly adsorbed ('fractionated plasma separation and adsorption' or FPSA). The purified plasma is then returned to the blood side of the albumin filter. In order to eliminate water-soluble toxins, blood thereafter undergoes hemodialysis using a conventional high-flux dialyser.

We hypothesise that removal of protein bound uremic retention solutes can be improved by FPSA as compared to standard hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* maintenance (> 3 months) hemodialysis patient
* Stable access, blood flow at least 250 mL/min

Exclusion Criteria:

* Known hemodialysis-related hypotension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2005-04; Study Completion 2009-12

PRIMARY OUTCOMES:
Uremic retention solute reduction rate
Biocompatibility

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Evenepoel, MD, Study Director — UZ Leuven; Kathleen Claes, MD, Principal Investigator — UZ Leuven; Björn Meijers, MD, Principal Investigator — UZ Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Vlaams-Brabant, Belgium